CLINICAL TRIAL: NCT05082233
Title: A Multicentre, Open-label, ph2 Clinical Study to Investigate the Efficacy, Safety, and Tolerance of Different Doses of Oral SHR7280 Tablets in Controlled Ovarian Hyperstimulation for Chinese Female Subjects Undergoing Assisted Reproductive Technology (ART)
Brief Title: Identify Effective Doses of SHR7280 Tablets in Controlled Ovarian Hyperstimulation (COH) for Female Subjects Undergoing Assisted Reproductive Technology (ART)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR7280-201
Record Dates: First submitted 2021-09-29; First posted 2021-10-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Female Subjects Undergoing COH in ART to Prevent Early Ovulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR7280 tablets (Experimental): Treatment group A: oral SHR7280 tablets; 300mg bid p.o.; Treatment group B: oral SHR7280 tablets; 200mg bid p.o.; Treatment group C: oral SHR7280 tablets; 200mg qd p.o.; Treatment group D: oral SHR7280 tablets; 400mg bid p.o.; as an alternative.
  Interventions: Drug: SHR7280 tablets

INTERVENTIONS:
Drug: SHR7280 tablets — Treatment group A:SHR7280 tablets ; 300mg BID； Treatment group B:SHR7280 tablets ; 200mg BID； Treatment group C:SHR7280 tablets ; 200mg QD； Treatment group D:SHR7280 tablets ; 400mg BID；

SUMMARY:
This study is a multicentre, open-label phase II dose-finding clinical trial that will recruit approximately 120 female subjects undergoing COH for in vitro fertilization (IVF) or intracytoplasmic single sperm injection (ICSI). We set up three SHR7280 tablets dose groups of 300 mg BID, 200 mg BID, and 200 mg QD with 40 subjects in each group, besides, a group of 400mg bid is set as an alternative.

ELIGIBILITY:
Inclusion Criteria:

1. Married infertile female subjects aged 20 to 39 years with indications for in vitro fertilization-embryo transfer (IVF-ET) or intracytoplasmic monosperm microinjection (ICSI) techniques.
2. Body mass index (BMI) of 18 to 28 kg/m2.
3. Regular menstrual cycle (24 to 35 days) for the last 3 months prior to screening.
4. Screening serum sex hormone levels must be performed on day 2 to 3 in the menstrual cycle and meet basal serum follicle stimulating hormone (FSH) < 10 IU/L; LH, estradiol (E2), progesterone (P), prolactin (PRL), and total testosterone levels within the normal laboratory range, or the investigator considers the abnormality without clinical significance; 1.2 ng/mL < anti-müllerian hormone (AMH) < 4.0 ng/mL.
5. Expected normal ovarian response.
6. Clinical feasible and willingness of the subject to undergo fresh cycle transfer with one or two embryos at a time in the first IVF-ET cycle.
7. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Subjects underwent 3 or more controlled ovarian stimulation cycles of IVF/ICSI-ET prior to screening without achieving clinical pregnancy.
2. Previous IVF or ART failure due to sperm/fertilization problems and no improvement in related medical condition.
3. Subjects had spontaneous abortion≥2 times.
4. Subjects at high risk of OHSS, judged by the investigator according to the Golan classification (e.g., those with moderate to severe OHSS during previous superovulatory cycles, polycystic ovary syndrome (PCOS) [refer to the 2018 Chinese PCOS guidelines] [1], or with previous cancelled cycles due to OHSS).

   Note: The 2018 Chinese PCOS guideline specifies the diagnostic criteria as meeting 1 of the following 2 items: ① hyperandrogenic manifestations or irregular menstruation: scanty or amenorrhea menstruation or irregular uterine bleeding are required for the diagnosis. ②Other diseases that may cause hyperandrogenism or abnormal ovulation should be excluded.
5. Subjects with low ovarian function meeting at least one of the following items: poor previous ovarian response (≤3 ovums obtained with previous conventional adequate Gn stimulation regimen); less than 7 follicles of 2-9 mm diameter (AFC) count visible on vaginal ultrasound in both ovaries; anti-mullerian hormone (AMH) < 1.1 ng/mL.
6. Any pregnancy that occurred within 3 months prior to screening date.
7. Subjects with clinically significant abnormal cervical findings within 6 months prior to screening (TCT).

   Note: Human papillomavirus (HPV) testing may be used as an adjunct in subjects with atypical squamous cells of undefined significance (ASC-US). Subjects may be included in the study if only the high-risk HPV strains test was negative.
8. Unexplained abnormal vaginal bleeding.
9. Persons who have donated blood or blood components within 1 month prior to screening, or have lost at least the equivalent of 200 mL of blood, or have received a blood transfusion within 2 months.
10. Subjects had a serious infection, severe trauma or major surgical procedure within 6 months prior to screening.
11. Use of clomiphene citrate, letrozole, gonadotropins (Gn), metformin, or oral contraceptives within 1 month prior to receiving ovarian stimulation.
12. Abnormal blood alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values on screening visit or ovarian stimulation day 1 visit.
13. Positive serum beta-hCG test result on day 1 of screening visit or ovarian stimulation.
14. Positive results for infectious diseases (including hepatitis B virus surface antigen, hepatitis C virus antibodies, human immunodeficiency virus antibodies, and syphilis spirochete antibodies).
15. Subjects with clinically significant abnormalities of the uterus and ovaries judged by the investigator, (e.g., submucosal fibroids, interstitial fibroids larger than 3 cm or less than 3 cm but affecting the morphology of the uterine cavity, untreated endometrial polyps, uterine adhesions, uterine malformations, ASRM stage III-IV endometriosis).
16. Any disease or condition that can affect the function of body systems and may affect the absorption, excessive accumulation, affect metabolism, or alter the excretion pattern of the study drug (e.g., chronic bowel disease, Crohn's disease, ulcerative colitis).
17. Subjects with clinically significant systemic disease, endocrine or metabolic abnormalities.
18. Previous or current thromboembolic disease.
19. Subjects or their spouses with structural chromosomal abnormalities, or with known monogenic genetic disorders or serious diseases with genetic susceptibility requiring preimplantation genetic testing (PGT).
20. History of tobacco or alcohol abuse within 3 months prior to screening: tobacco addiction (more than 5 cigarettes or equivalent per day); alcohol abuse (greater or equal to 14 units of alcohol per week: 1 unit = 360 mL of beer, or 25 mL of spirits 40% or more in strength, or 1 glass of wine, 180 mL).
21. History of substance abuse, drug dependence.
22. Allergy or allergy to two or more foods or drugs, including known history of allergy to the study drug or any component of the study drug.
23. Subjects that have participated in a clinical trial of any drug or medical device within 3 months prior to screening, or are still within the follow-up period of a clinical study or within 5 half-lives of the trial drug (depends on the longer one) prior to screening
24. History of malignant tumors of the ovaries, breast, uterus, hypothalamus, pituitary gland, etc.
25. Subjects with serious mental disease or who are unable to understand the purpose and methods of this clinical trial.
26. Any other reason deemed by the investigator to be unsuitable for participation in this study.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Inhibition rate of early LH serge with different oral doses of SHR7280 tablets from the 1st day of study drug administration to the date of hCG injection | Through the whole period of oral administration of SHR7280, generally 5-7 days)

SECONDARY OUTCOMES:
The proportion of embryos with 2 protoplasts in the cytoplasm 16-18 hours (h) after fertilization (2PN rates). | On embryo transfer day, 3 days after oocyte retrieval
Quality embryo rates | On embryo transfer day, 3 days after oocyte retrieval.
Clinical pregnancy rates. | On pregnancy test day
Total dose of gonadotropin (Gn) administered and duration of gonadotropin treatment | Through the whole period of controlled ovarian stimulation, generally 9-11 days
Adverse drug events | Through study completion, follow-up period may be up to 40 weeks if the patient gets a successful clinical pregnancy and a full term delivery
Population PK endpoints: analysis of plasma SHR7280 concentration data, population pharmacokinetic modeling, and calculation of key pharmacokinetic parameters of SHR7280 in subjects | Blood samples were collected within 30 minutes before,, 1-3 hours after and 5-8 hours after the oral administration of SHR7280 in the morning on hCG injection day, generally the 9th day to the 11st day of the period of controlled ovarian stimulation
PD endpoints: serum E2, luteinizing hormone (LH) and progesterone (P) concentrations at each time point | 30 minutes before the oral administration of SHR7280 every morning during SHR7280 treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chi H, Song Y, Jin L, Song X, Wang X, Ma Q, Cao Y, Liang X, Tan J, Guan Y, Diao F, Li Y, Li Z, Sun Y, Shu C, Chen H, Shen K, Qiao J. SHR7280, an oral gonadotropin-releasing hormone antagonist, for the prevention of premature luteinizing hormone surge in controlled ovarian hyperstimulation: a dose-finding, phase 2 trial. Hum Reprod. 2025 Jul 1;40(7):1357-1365. doi: 10.1093/humrep/deaf082. PMID 40373184